CLINICAL TRIAL: NCT06329752
Title: Ultrasound-guided Sciatic Nerve Block for Distal Leg and Ankle Fracture Manipulation in the Emergency Department: A Feasibility Study
Brief Title: Sciatic Nerve Block for Ankle and Leg Fracture Manipulation in the Emergency Department
Acronym: AnkleMan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Santi Di Pietro, Emergency Medicine Consultant, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Not available yet
Record Dates: First submitted 2024-02-20; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Ankle Fractures; Leg Fracture
MeSH Terms: conditions — Ankle Fractures | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Interventional, single-arm, feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sciatic Nerve block Arm (Single Arm) (Experimental)
  Interventions: Procedure: Ultrasound-guided Sciatic Nerve block (20 mL of 2% Lidocaine)

INTERVENTIONS:
Procedure: Ultrasound-guided Sciatic Nerve block (20 mL of 2% Lidocaine) — Patients will be scanned with the ultrasound machine to determine the technical feasibility of sciatic nerve blocks. If feasible, one of the following techniques will be performed a) popliteal sciatic nerve block, with either lateral or posterior approach; b) CAPS (crosswise approach to popliteal sciatic) block, with either lateral to medial or anterolateral to posteromedial approach; c) subgluteal sciatic nerve block; d) transgluteal sciatic nerve block. In all cases, 20 mL of 2% Lidocaine will be used.

SUMMARY:
The goal of this feasibility clinical trial is to assess the acceptability of ultrasound-guided sciatic nerve block when performed at Emergency Departments for manipulation and temporary stabilization of distal leg and ankle fractures.

The trial aims to assess:

* The acceptability of sciatic nerve block
* The technical feasibility of sciatic nerve block
* The technical success of sciatic nerve block
* The analgesic efficacy of sciatic nerve block

In addition to that, this study aims to

* Describe patient-reported and physician-reported satisfaction
* Assess the Adverse Event rate at 48 hours post intervention

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Confirmed radiological diagnosis of distal tibia fracture (Group 43 according to AO classification, all subtypes included); or malleolar fracture (Group 44 according to AO classification, all subtypes included); or distal fibula fracture (Group 4F3 according to AO classification, both the two subtypes included); or any combination of the fracture patterns described
* Fractures requiring manipulation in the ED to achieve temporary stabilization either as manual reduction and cast immobilization; or calcaneal pin traction (as per local policy or treating physician's preference)
* Capacity to understand the aim of the study, the potential benefits and harms of the proposed intervention
* Capacity to provide consent
* Capacity to provide a self-assessment of pain using the written VAS Scale

Exclusion Criteria:

* Fractures that do not require any form of manipulation in the ED according to the treating physician (e.g., fractures with minimal or no displacement of the bony fragments, that are immobilized in a posterior leg cast by the nursing stuff/physicians assistants without any painful manipulations of the bony fragments performed by the physician)
* Open fractures
* Perisynthetic or periprosthetic fractures
* Distal leg/ankle fractures with neurovascular compromise
* Clinical signs of compartment syndrome
* Skin infection at the needle entry sites
* Diabetic neuropathy or any other known form of neuropathy that causes reduced sensation in the sciatic and/or femoral nerve territory
* Charcot-Marie-Tooth disease
* Known allergy to local anaesthetics or opioids
* Hemodynamic instability
* Known diagnosis of severe cognitive impairment
* Dementia and/or delirium (defined by a 4AT score ≥ 2)
* Lack of capacity to provide consent and to understand the aim of the study
* Patient's refusal to participate in the study
* BMI>35
* Body weight < 40 Kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
To assess the technical feasibility of ultrasound-guided sciatic nerve block when performed at Emergency Departments for manipulation and temporary stabilization of distal leg and ankle fractures. | From patient recruitment until sciatic nerve scanning (an estimated time frame of 30 minutes)
  Percentage of patients for whom the block is deemed technically feasible by the investigator in charge of this task

SECONDARY OUTCOMES:
Technical success of US-guided sciatic nerve block | 15 Minutes post US-guided sciatic nerve block
  Percentage of patients treated with sciatic nerve block who develop complete or mild- score 0 or 1 - sensory deficit 15 minutes post block
Analgesic efficacy of US-guided sciatic nerve block | An estimated average time of 15 minutes after the beginning of fracture manipulation
  Percentage of patients manipulated after a successful sciatic nerve block who report Pain Max < 40 mm
Patient-reported and physician-reported satisfaction | An estimated average time of 30 minutes after the beginning of fracture manipulation
  Patient's satisfaction and Treating physician's satisfaction assessed with a 5-points Likert scale.

OTHER OUTCOMES:
Safety Endpoint | In the first 48 hours post intervention
  Number and type of adverse events in the first 48 hours post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Santi Di Pietro, MD, Principal Investigator — University of Pavia - IRCCS San Matteo University Hospital
Locations (1):
- Emergency Department, IRCCS Fondazione Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No